CLINICAL TRIAL: NCT05366166
Title: A Phase II Trial of Induction and Maintenance Pembrolizumab and Olaparib in Locally Advanced Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Pembrolizumab Plus Olaparib in LA-HNSCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2047
Record Dates: First submitted 2022-05-04; First posted 2022-05-09 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: head and neck; squamous cell carcinoma; HPV negative; pembrolizumab; olaparib; PARP inhibitor; anti-PD1 inhibitor; intensity modulation radiation therapy; Proton therapy; cisplatin
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — pembrolizumab; olaparib; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): The participants will receive neoadjuvant and adjuvant pembrolizumab and olaparib combination plus standard of care (chemoradiation therapy) as defined in the protocol.
  Interventions: Biological: Pembrolizumab; Drug: Olaparib; Drug: Cisplatin; Radiation: IMRT (intensity modulated radiation therapy)

INTERVENTIONS:
Biological: Pembrolizumab — In the induction phase, participants will receive a single intravenous infusion of pembrolizumab 400 mg prior to chemoradiotherapy. In the Maintenance Phase, participants will receive pembrolizumab 400 mg every 42 days for 8 cycles.
  Other Names: KEYTRUDA®; MK-3475
Drug: Olaparib — In the induction phase, participants will receive daily oral olaparib 150 mg two times a day for 3 weeks prior to chemoradiotherapy. In the Maintenance Phase, participants will receive daily olaparib 150 mg two times a day for up to 48 weeks.
  Other Names: AZD-2281; MK-7339; KU0059436
Drug: Cisplatin — In the chemoradiation phase, participants will receive weekly intravenous cisplatin infusion, 40 mg/m2 over 7 weeks.
  In the chemoradiation phase, standard of care radiation therapy and chemotherapy will be administered, for a total of 7 weeks. Radiation therapy is done on daily basis (excluding weekends), and chemotherapy therapy will involve cisplatin infusion once weekly.
  Other Names: CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-platinum
Radiation: IMRT (intensity modulated radiation therapy) — In the chemoradiation phase, participants will receive 70 Gray external beam radiotherapy, at 2 Gray/fraction dose, 35 fractions, delivered once a day, on weekdays, using Intensity Modulated Radiotherapy Treatments or proton radiotherapy techniques, over 7 weeks.

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of using a combination of pembrolizumab and olaparib when given before and after standard chemoradiation therapy in treating locally advanced head and neck squamous cell carcinoma. Pembrolizumab and olaparib are drugs that are approved for head and neck cancer treatment. However, FDA has not approved the use of these two drugs together in treating head and neck cancer.

DETAILED DESCRIPTION:
Treatment outcomes are poor for patients with locally advance human papilloma virus (HPV) negative and high-risk HPV positive head and neck squamous cell carcinoma (HNSCC). One standard of care (SOC) for HNSCC is definitive chemoradiotherapy (CRT). This study will evaluate the safety and efficacy of the addition of pembrolizumab, an anti-programmed death-1 (PD1) inhibitor, and olaparib, a Polyadenosine 5'diphosphoribose polymerization (PARP) inhibitor, before and after SOC CRT, which will be delivered in 70 Gray in 35 fractions with concurrent weekly cisplatin 40 mg/m2 over 7 weeks.

Treatment will be offered in three sequential phases. In the induction phase, participants will receive one infusion of pembrolizumab and will take olaparib tablets for a total of 21 days. In the chemoradiation phase, radiation therapy will administered daily (excluding weekends) and cisplatin infusion will be given weekly. In the maintenance phase, pembrolizumab infusion will be done once every 6 weeks in additional to twice daily olaparib tablets for up to 8 treatment cycles that are 42-days per cycle.

ELIGIBILITY:
Inclusion Criteria:

In order to participate in this study, a subject must meet all of the eligibility criteria outlined below.

1. Age >18 years on the day of signing the consent
2. Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
3. Subject is willing and able to comply with study procedures based on the judgment of the investigator or protocol designee. The subject must be willing to consent to a mandatory pre-study biopsy unless sufficient archival tissue is available.
4. Biopsy confirmed American Joint Committee on Cancer 8th Edition35 stage III-IV B oral cavity squamous cell carcinoma (SCC), p16-negative oropharyngeal SCC, stage III-IVB hypopharyngeal SCC, stage III-IVB laryngeal SCC -OR- HPV-associated oropharyngeal SCC (p16 positive or HPV-associated) T4 or N3 , T1-3 N2 or T3N0-1 with >10 pack-year tobacco history
5. At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by imaging (CT/ PET) and is suitable for repeated assessment.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. No prior curative attempts for this cancer (i.e., surgery, radiation, systemic therapy) and not currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of the study intervention. No evidence of metastatic disease (M0)

Exclusion Criteria

1. Subjects with prior and concurrent malignancies of different tumor types whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the study drug are eligible with the following exception: Subjects with prior history of HNSCC treated < 3 years to the date of consent.
2. Cisplatin-ineligible as defined in the protocol.
3. Severe, active medical comorbidity. Subjects are considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography scan or any psychiatric disorder that prohibits obtaining informed consent.
4. Subjects unable to swallow orally administered medication prior to initiation of study treatment.
5. Systemic glucocorticoids for any purpose other than to modulate symptoms from an event of clinical interest of suspected immunologic etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2030-11-21 (Estimated)

PRIMARY OUTCOMES:
One Year Progression Free Survival (PFS) | up to 1 year from start of treatment
  One Year PFS will be defined as the period from the date of treatment start until disease progression or death (whichever occurs first) up to one year. Subjects who have not had an event will be censored at the date of last disease assessment documenting the subject was free of progression. Progression will be evaluated by RECIST v1.1
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Overall survival | up to 2 years from start of treatment
  Overall survival will be defined as the period from the date of treatment start until death of any cause. Subjects who have not had an event will be censored at the date of last assessment documenting the subject was alive.
Two Year Progression Free Survival (PFS) | Up to 2 years from start of treatment
  Two Year PFS will be defined as the period from the date of treatment start until disease progression or death (whichever occurs first) up to two year. Subjects who have not had an event will be censored at the date of last disease assessment documenting the subject was free of progression. Progression will be evaluated by RECIST v1.1
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Induction therapy related delays in chemoradiation therapy | Up to 14 weeks from start of treatment
  Induction therapy related delays in chemoradiation therapy (CRT) will be defined type and associated grade of toxicity according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0. criteria and days of delay to start CRT due to induction one cycle of induction pembrolizumab and olaparib.
Toxicities related to maintenance therapy | Up to 2 years from start of treatment
  Toxicities related to maintenance therapy associated with pembrolizumab and olaparib will be classified and graded according to NCI-CTCAE v5.0.
  The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Induction related toxicity using patient-reported outcomes | Up to 2 years from start of treatment
  Induction pembrolizumab and olaparib related toxicity will be defined using Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) in subjects receiving one cycle of pembrolizumab and olaparib.
Patient reported maintenance therapy-related toxicities | Up to 2 years from start of treatment
  Maintenance therapy-related toxicities using patient-reported outcomes (PRO-CTCAE) in subjects who received induction pembrolizumab with olaparib, followed by definitive treatment with concurrent cisplatin-radiotherapy and maintenance pembrolizumab and olaparib.
One-year locoregional control | Up to 1 year from start of treatment
  One-year locoregional control will be defined as the period from the start of treatment until recurrence at primary site or nodal site (whichever occurs first) as defined by RECIST 1.1
Distant Metastasis-Free Survival (DMFS) | Up to 1 year from start of treatment
  DMFS will be defined as the period from the date of treatment start until distant metastasis or death (whichever occurs first) as defined by RECIST 1.1. Subjects who have not had an event will be censored at the date of last disease assessment documenting the subject was free of distant metastasis.
Correlate Combined Positive Score (CPS) and one-year progression free survival (PFS) | Up to 1 year
  To correlate combined positive score (CPS) with one-year PFS, quality of life scores will be summarized using descriptive statistics like mean, sd, median, range, in participants who received induction pembrolizumab with olaparib, followed by definitive treatment with concurrent cisplatin-radiotherapy and maintenance pembrolizumab and olaparib.
Head and Neck Cancer Associated Patient Reported Outcomes (PRO) | Baseline, 4week, 7 week, 12 weeks, 6months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  Head and Neck Cancer Associated PRO will be evaluated using European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Head and Neck Module (QLQ-H&N35).
  EORTC QLQ-H&N35 has 35 questions assessing symptoms and side effects of treatment, social function and body image/sexuality. Most questions used 4 point scale (1 'Not at all' to 4 'Very much'); several single item questions were just coded as no=1, yes=2. The scores transformed and analyzed on a 0 - 100 scale. High scores indicate more problems.
General Cancer Associated Patient Reported Outcomes (PRO) | Baseline, 4week, 7week, 12 weeks, 6 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months
  General Cancer Associated PRO will be evaluated using European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ-C30).
  The EORTC QLQ-C30 has 30 questions, 9 multi-items: 5 functional, 9 symptoms and a global health and quality-of-life. Most questions used 4-point scale (1 'Not at all' to 4 'Very much'); 2 questions used 7-point scale (1 'very poor' to 7 'Excellent'). The scores transformed and analyzed on a 0 - 100 scale. A higher score=better.

CONTACTS AND LOCATIONS:
Overall Officials: Siddharth Sheth, DO MPH, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (4):
- United States (4):
  - Indiana University Simon Comprehensive Cancer Center, Indianapolis, Indiana
  - University of Louisville, Brown Cancer Center, Louisville, Kentucky
  - UNC Lineberger, Chapel Hill, North Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials